CLINICAL TRIAL: NCT02223611
Title: Phase ⅡTrial of S1 Capsule Plus Cisplatin Versus Vinorelbine Plus Cisplatin as Adjuvant Treatment in Stage Ⅱ-ⅢA Non-small Cell Lung Cancer (NSCLC) After Complete Resection
Brief Title: Clinical Observation of S1 Capsule for Stage Ⅱ-ⅢA Non-small Cell Lung Cancer After Complete Resection
Acronym: S1VSNP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HBMF9990
Record Dates: First submitted 2014-08-14; First posted 2014-08-22 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Non-small Cell Lung Cancer Stage Ⅱ; Non-small Cell Lung Cancer Stage ⅢA
Keywords: Stage Ⅱ-ⅢA NSCLC S1 capsule Completely resection
MeSH Terms: interventions — S 1 (combination); Cisplatin; Injections; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- S1 capsule plus Cisplatin (Experimental): S1: 40mg, bid, when body surface area (BSA)<1.25 m2, 50mg; bid when 1.25 m2≤BSA<1.5 m2; 60mg, bid when 1.5 m2≤BSA 60mg from day 1 to 14. Cisplatin: 75 mg/m2 on day 1.
  3 weeks/4cycles
  Interventions: Drug: S1 capsule
- Vinorelbine plus Cisplatin (Active Comparator): Vinorelbine: 25 mg/m2 intravenously on day 1, and day 8. Cisplatin: 75 mg/m2 intravenously on day 1.
  3 weeks/4cycles
  Interventions: Drug: Vinorelbine

INTERVENTIONS:
Drug: S1 capsule — Within four weeks after the completely resection, S-1 was administered orally twice a day, after meals on days 1 to 14. The actual dose of S-1 was selected as follows: in a patient with body surface area (BSA)<1.25 m2 40mg twice a day, 1.25 m2≤BSA<1.5 m2 50mg twice a day, and 1.5 m2≤BSA 60mg twice a day. Cisplatin (75 mg/m2) was administered intravenously on day 1 The treatment regimen was repeated every 3 weeks, totally 4 cycles unless disease progression or unacceptable toxicity occurred.
  Other Names: S1: Gimeracil and oteracil porassium capsules; Cisplatin: Cisplatin for injection
  Arms: S1 capsule plus Cisplatin
Drug: Vinorelbine — Vinorelbine (25 mg/m2) is administered intravenously on day 1, and day 8. Cisplatin (75 mg/m2) is administered intravenously on day 1. The treatment regimen is repeated every 3 weeks, totally 4 cycles unless disease progression or unacceptable toxicity occurred.
  Other Names: Vinorelbine: Navelbine,vinorelbine bitartrate injection; Cisplatin: Cisplatin for injection
  Arms: Vinorelbine plus Cisplatin

SUMMARY:
The purpose of this study is to evaluate S1 capsule plus Cisplatin as adjuvant treatment in stageⅡ and Ⅲa non-small cell lung cancer. It is the first study in the world to investigate the safety and efficacy of S1 capsule using in stageⅡ and Ⅲa non-small cell lung cancer patients after the complete resection.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer death worldwide. Only about 15.6% of all lung cancer patients are alive 5years or more after diagnosis. Non-small Cell Lung Cancer (NSCLC) accounts for more than 85% of all lung cancer cases.

For individuals with stage Ⅱ-ⅢA NSCLC after complete resection, platinum-based chemotherapy is the mainstay of first line treatment. Various treatment regimens have been developed to improve survival.

S-1 capsule is an novel oral anticancer drug that combines tegafur, a prodrug of 5-fluorouracil, with gimeracil and oteracil potassium. S-1 capsule was considered to be an active single agent against NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Patient with completely resected stage ⅢA non-small cell lung cancer(NSCLC)
* Must be able to receive the therapy of the study within four weeks after the completely resection

Exclusion Criteria:

* Systemic anticancer treatment
* local radiotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Disease free survival rate | 2 years

SECONDARY OUTCOMES:
Disease free survival | 4 years
  The period from the date of enrollment to the date on which the recurrence was first confirmed. For patients who died before disease progression from any cause, death was attributed to recurrence.
Overall survival | 4 years
  The period from the date of enrollment to the date of death from any cause.
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Participants will be followed for the duration of hospital stay, an expected average of 3 weeks.
  The incidences of adverse events were calculated according to the National Cancer Institute Cancer Common Toxicity Criteria, version 4.0.
Quality of life (QOL) | Participants will be followed for the duration of hospital stay, an expected average of 3 weeks.
  QOL was assessed with the lung cancer subscale of the Functional Assessment of Cancer Therapy-Lung (FACT-L) and Lung Cancer Symptom Scale(LCSS).

OTHER OUTCOMES:
Molecular marker measurement for NSCLC | Some molecular markers in the serum will be tested at 6-month intervals after surgery until recurrence
  The measured molecular markers include carcinoembryonic antigen (CEA), tissue polypeptide specific antigen (TPS), neuron-specific enolase (NSE), carbohydrate antigen 199 (CA199), cytokeratin fragment 19 ( CYFRA 21-1), and squamous cell carcinoma antigen (SCC Ag)

CONTACTS AND LOCATIONS:
Overall Officials: Jun-Feng Liu, Professor, Principal Investigator — Department of Thoracic Surgery Fourth Hospital, Hebei Medical University, China
Locations (1):
- Jun Feng Liu, Shijiazhuang, Hebei, China